CLINICAL TRIAL: NCT03608189
Title: Multimodal Assessment of Knee Conditions in Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Other Study IDs: 24302214-1; 24302214 (Other: University of Oulu)
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: ACL Injury
Keywords: Osteoarthritis; ACL injury; Knee trauma; Meniscus tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACL injury subjects: Subjects with anterior cruciate ligament injuries.

SUMMARY:
The purpose of this study is to assess ACL injury and other pathological knee conditions from the combination of signals that are known to provide information on the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* ACL injury
* Ages 18-40
* Female

Exclusion Criteria:

* BMI under 18
* BMI over 40
* Contraindications to MRI

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient participating in rehabilitation due to ACL injuries and potential other knee disorders.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective evaluation method for knee disorder recovery | Six months
  ACL injury recovery (confirmed by using MRI)

CONTACTS AND LOCATIONS:
Overall Officials: Simo Saarakkala, Ph.D., Principal Investigator — University of Oulu; Osmo Tervonen, Ph.D., M.D., Study Director — Oulu University Hospital
Locations (1):
- University of Oulu, Oulu, North Ostrobothnia, Finland

IPD SHARING:
Plan to Share IPD: Undecided